CLINICAL TRIAL: NCT05136703
Title: Treatment Research Investigating Depression Effects on Neuroimmune Targets (TRIDENT)
Acronym: TRIDENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Adam Carrico, PhD, Professor, Florida International University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 20210773; R01MH128868 (NIH)
Record Dates: First submitted 2021-11-15; First posted 2021-11-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Depression; HIV-1-infection; Inflammation
Keywords: Depression; Microbiome; HIV; CBT-AD; Gut; Brain
MeSH Terms: conditions — Depression; Inflammation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-Behavioral Therapy for Adherence and Depression (CBT-AD) (Experimental): Participants randomized to receive CBT-AD immediately will complete up to 15 individual sessions (12 session with 3 booster sessions) focused on depression and one session of ART Adherence counseling during the four months following randomization.
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Adherence and Depression (CBT-AD); Behavioral: Antiretroviral Therapy (ART) Adherence Counseling
- Wait-List Control (WLC) (Experimental): Participants randomized to the WLC condition will receive one session of ART adherence counseling immediately following randomization. After six months, WLC participants will have the opportunity to receive 15 individually delivered CBT-AD sessions (12 sessions and 3 booster sessions) focused on depression.
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Adherence and Depression (CBT-AD); Behavioral: Antiretroviral Therapy (ART) Adherence Counseling

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy for Adherence and Depression (CBT-AD) — CBT-AD is a behavioral intervention administered either in person or via Zoom. Each session lasts approximately 50 minutes. Participants will receive up to 12 individually delivered sessions over 4 months. Participants receive up to three individually delivered booster sessions through 6 months.
Behavioral: Antiretroviral Therapy (ART) Adherence Counseling — This treatment involves a single session integrating CBT for depression with CBT for adherence following our "Life-Steps" approach.

SUMMARY:
The purpose of this randomized controlled trial is to understand how a cognitive-behavioral treatment (a form of psychological treatment) for depression changes the gut microbiome (micro-organisms that regulate the health of the gut), immune system, and the brain functioning in people living with HIV.

DETAILED DESCRIPTION:
The overarching goal of this randomized controlled trial (RCT) is to identify the causal pathways that drive depressive symptoms among people with HIV (PWH). The scientific premise is that evidence-based depression treatment is an innovative, experimental probe to determine the neural substrates of depression and mechanistic relevance of microbiome-gut-brain (MGB) axis changes during and after Cognitive-Behavioral Therapy for Adherence and Depression (CBT-AD) on brain and behavioral function. The proposed causal pathway is that reductions in depressive symptoms following the delivery of CBT-AD treatment will trigger a cascade of alterations in the MGB axis. Specifically, CBT-AD related decreases in depressive symptoms will induce alterations in gut dysbiosis, decrease microbial translocation, and improve soluble neuroactive markers of peripheral immune dysregulation. Our efforts to elucidate the immunologic mechanisms whereby CBT-AD could improve neurobehavioral outcomes will also focus on an established leukocyte signaling pathway, the Conserved Transcriptional Response to Adversity (CTRA), which has been shown to be responsive to behavioral interventions and psychosocial factors outside of HIV.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Speaks and reads English
3. Verified HIV+ status with antiretroviral medications bearing his/her name
4. Current diagnosis on Major Depressive Disorder (MDD) using a structured clinical interview (DIAMOND) or Hamilton Rating Scale for Depression scores of 7 or greater
5. If prescribed antidepressants, on a stable regimen and dose for at least 2 months
6. Suppressed HIV viral load (< 200 copies/mL)
7. Able to complete Functional Magnetic Resonance Imaging (fMRI) scans (i.e., no claustrophobia, no metal implants, no pacemaker, and BMI < 40)

Exclusion Criteria:

1. Unable to provide informed consent
2. Active, untreated major mental illness
3. Pregnancy at baseline
4. Received CBT for depression in the past 2 years
5. 5. Otherwise eligible but does not complete the run-in period that includes the baseline assessment, biospecimen collection, the fMRI visit, and a separately scheduled randomization visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in resting state activation of the negative valence system | 6 Months
  Measured by functional Magnetic Resonance Imaging (fMRI)
Change in connectivity of the negative valence system | 6 Months
  Measured by functional Magnetic Resonance Imaging (fMRI)

SECONDARY OUTCOMES:
Depressive Symptoms | 6 Months
  The Hamilton Rating Scale for Depression is an interviewer-administered measure that has a total score ranging from 0-52 with the higher score indicating greater depressive symptoms
Alterations in gut microbiota | 4 months
  Measured via 16s sequencing of the gut microbiome using rectal swabs and fecal samples
Conserved transcriptional response to adversity (CTRA) leukocyte signaling pathway | 4 Months
  Measured using Ribonucleic Acid (RNA) sequencing from peripheral blood mononuclear cells
Soluble Markers of Microbial Translocation | 4 Months
  Enzyme-linked immunosorbent assay (ELISA) methods will be employed to measure lipopolysaccharide binding protein (LBP) levels in plasma samples. Log10 will be the unit of measure.
Soluble Markers of Immune Activation and Inflammation | 4 Months
  Enzyme-linked immunosorbent assay (ELISA) methods will be employed to measure levels of monocyte activation markers (i.e., soluble CD14, soluble CD163) and pro-inflammatory cytokines (e.g., interleukin, high sensitivity c-reactive protein) in plasma samples. Log10 will be the unit of measure.
Soluble Markers of Dysregulated Neurotransmitter Synthesis | 4 Months
  High performance liquid chromatography method with fluorescence will measure mean levels of the kynurenine/tryptophan and phenylalanine/tyrosine ratios in plasma samples. Log10 will be the unit of measure.
Neurocognitive Functioning | 6 Months
  Changes in mean levels of measures indexing executive functioning, attention, and affect regulation assessed in a comprehensive, interviewer-administered neuropsychological assessment battery. Units will be expressed as standardized scores (i.e., T scores).

CONTACTS AND LOCATIONS:
Overall Officials: Adam W Carrico, PhD, Principal Investigator — Florida International University
Locations (2):
- United States (2):
  - University of Miami Neuroimaging Facility, Coral Gables, Florida
  - Care Resource - Midtown Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: No